CLINICAL TRIAL: NCT03529708
Title: Stereotactic Body Radiotherapy (SBRT) Boost Following Urgent 3D Conformal Radiotherapy in the Treatment of Metastatic Epidural Spinal Cord Compression (SCC): A Phase I Feasibility Trial
Brief Title: Stereotactic Body Radiotherapy Boost After Palliative Radiotherapy for Spinal Cord Compression
Acronym: CRUSSH
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Juravinski Cancer Center (Other)
Collaborators: Hamilton Health Sciences Corporation (Other); Juravinski Cancer Centre Foundation (Other)
Responsible Party: Principal Investigator, Elysia Donovan, Elysia Donovan, MD FRCPC, Radiation Oncology, McMaster University, Juravinski Cancer Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 4760
Record Dates: First submitted 2018-04-24; First posted 2018-05-18 (Actual); Last update posted 2020-01-29 (Actual); Status verified 2020-01

CONDITIONS: Spinal Cord Compression; Cauda Equina Syndrome; Stereotactic Body Radiotherapy
MeSH Terms: conditions — Spinal Cord Compression; Cauda Equina Syndrome | interventions — Radiotherapy, Conformal

STUDY DESIGN:
Intervention Model Description: Single arm pilot study of standard of care 3D conformal radiotherapy plus Stereotactic body radiotherapy (SBRT) boost
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- SBRT boost (Experimental): Standard radiotherapy (3D conformal, urgent palliative radiotherapy) plus stereotactic body radiotherapy (SBRT) boost
  Interventions: Radiation: 3D CRT plus SBRT boost

INTERVENTIONS:
Radiation: 3D CRT plus SBRT boost — Patients will receive urgent standard 3D conformal radiotherapy (3D CRT) of plus stereotactic boost to tumor causing spinal cord compression (SCC). Initial dose for 3D CRT will be either 8Gy in 1 fraction or 20Gy in 5 fractions, with SBRT boost dose15Gy in 2 fractions of 12Gy in 2 fractions (depending on 8Gy/1 or 20Gy/5 initial RT dose respectively), delivered within three weeks of first treatment.

SUMMARY:
Spinal cord compression (SCC) is a devastating complication of advanced malignancy, and can cause significant deterioration in function and quality of life (QoL). The goal of treatment is to improve functional status and symptoms, but the optimal treatment regimen for these patients has not been thoroughly established. Many patients with SCC present with uncontrolled systemic disease and poor performance status, and are not eligible for standard surgical resection. They are generally treated with 3D conformal palliative RT (3DCRT) alone, however recent trials suggest that less than 70% of patients are ambulatory, that the re-establishment of ambulation in non-ambulatory patients is poor, and the duration of improvement is guarded with radiotherapy alone.

Recently, stereotactic body radiotherapy (SBRT) used alone or after previous radiotherapy to treat spinal metastasis has demonstrated superior results in pain control, tumour response and durability. SBRT requires time for careful planning, and many patients with neurologic symptoms must be treated immediately to prevent progression. Therefore the role of SBRT is still unclear in this patient population, although it seems to be a potential alternative to surgical decompression in patient not suitable for surgery. The investigators propose a feasibility study to investigate the potential benefits of dose escalation with a sequential SBRT boost to urgent 3D CRT in the setting of SCC. This regimen will allow inoperable patients to receive urgent 3DCRT while simultaneously creating the opportunity for superior outcomes with SBRT. The investigators also aim to characterize the effect on motor function and ambulation, pain and QoL. This study could stimulate further multi-center randomized trials in this area, improve motor function and patient-reported QoL, and contribute to improving oncology care in Canada in a meaningful way.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of metastatic malignancy (radiologic or pathologic)
2. Evidence of disease in vertebral body with epidural component such that Bilsky radiologic score is 1c-2 on MRI (abuts spinal cord without cord compression (1c), or spinal cord compression but with visible CSF (2)
3. Motor function (MF) of 3 or greater

Exclusion Criteria:

1. Surgical candidate
2. Instability of vertebral bodies with or without bony retropulsion requiring surgical intervention or hardware placement
3. Previous radiotherapy course to same region of spine with overlapping fields (prior to phase I course) at discretion of treating radiation oncologist
4. No CT or MRI within previous 3 months
5. Life expectancy estimated <3 months
6. Performance status KPS<40
7. On active chemotherapy or targeted therapy or immunotherapy (must be stopped for at least one week prior to and following)
8. Pregnant or lactating
9. Contraindications to radiotherapy (eg. active autoimmune disease requiring medication)
10. Inability to lie flat comfortably for at least 20 minutes
11. Age < 18

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2018-06-01 (Actual); Primary Completion 2020-06-01 (Estimated); Study Completion 2020-12-01 (Estimated)

PRIMARY OUTCOMES:
Feasibility of accrual | up to 12 months
  Success determined by accrual of 30 patients with SBRT boost is planned and delivered to 80% of these

SECONDARY OUTCOMES:
Motor Function Description: | 4 weeks (primary), 12 weeks, 6 months
  Motor strength evaluated by 8 point scale (0= Complete paraplegia, 1= Palpable or visible muscle contractions, 2= Active movement of the leg without gravity, 3= Active movement of the leg against gravity, 4= Active movement againt mild resistance, 5= Active movement against intermediate resistance, 6= Active movement against strong resistance, 7= Normal strength)
Overall Quality of Life (QoL) | 4 weeks, 12 weeks, 6 months
  Change in total QoL score over time per European Organization for Research and Treatment of Cancer Quality of Life Questionnaire core 30 (EORTC QLQ-c30)
Pain Response | 4 weeks, 12 weeks, 6 months
  Change in level of pain over time on 10 point scale with 0 meaning no pain and 10 meaning severe pain (patient-reported)
Local Control | 12 weeks, 6 months
  Assessment of tumor volume (maximum size in 3 dimension) by Magnetic Resonance Imaging (MRI)
Toxicity | 4 weeks, 12 weeks, 6 months
  Treatment-related toxicity graded by Common Terminology for Adverse Events (CTCAE 4.03)
Overall Survival | 4 weeks, 12 weeks, 6 months
  Survival time from first radiotherapy treatment (3D CRT) in days
Bone metastasis- specific Quality of Life | 4 weeks, 12 weeks, 6 months
  Change in total QoL score over time per European Organization for Research and Treatment of Cancer Quality of Life Questionnaire Bone Metastasis-22 (EORTC QLQ BM-22)

CONTACTS AND LOCATIONS:
Locations (1):
- Juravinski Cancer Center, Hamilton, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Donovan EK, Greenspoon J, Schnarr KL, Whelan TJ, Wright JR, Hann C, Whitton A, Chow T, Parpia S, Swaminath A. A pilot study of stereotactic boost for malignant epidural spinal cord compression: clinical significance and initial dosimetric evaluation. Radiat Oncol. 2020 Nov 18;15(1):267. doi: 10.1186/s13014-020-01710-4. PMID 33208170